CLINICAL TRIAL: NCT07166419
Title: Phase I Clinical Trial of Caring Cross Anti-CD19/20/22 Chimeric Antigen Receptor T Cells for Treatment of Relapsed or Refractory Lymphoid Malignancies (Non-Hodgkin Lymphoma, Acute Lymphoblastic Leukemia, Chronic Lymphocytic Leukemia) (C3PO)
Brief Title: Anti-CD19/20/22 Chimeric Antigen Receptor T Cells (TriCAR19.20.22 T Cells) for the Treatment of Relapsed or Refractory Non-Hodgkin Lymphoma, Acute Lymphoblastic Leukemia, and Chronic Lymphocytic Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Sumithira Vasu, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-24176; NCI-2025-05721 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Blast Phase Chronic Myeloid Leukemia, BCR-ABL1 Positive; Recurrent Acute Lymphoblastic Leukemia; Recurrent Chronic Lymphocytic Leukemia; Recurrent Chronic Myeloid Leukemia, BCR-ABL1 Positive; Recurrent Indolent Non-Hodgkin Lymphoma; Recurrent Lymphoblastic Lymphoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Transformed Chronic Lymphocytic Leukemia; Refractory Acute Lymphoblastic Leukemia; Refractory Chronic Lymphocytic Leukemia; Refractory Chronic Myeloid Leukemia, BCR-ABL1 Positive; Refractory Indolent Non-Hodgkin Lymphoma; Refractory Lymphoblastic Lymphoma; Refractory Non-Hodgkin Lymphoma; Refractory Transformed Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Non-Hodgkin | interventions — Specimen Handling; Biopsy; Cyclophosphamide; fludarabine; Blood Component Removal; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (TriCAR19.20.22 T cells) (Experimental): Patients undergo apheresis between days -30 and -7 or days -9 and -7. Patients receive lymphodepletion chemotherapy with cyclophosphamide IV on day -6, fludarabine IV over 30 minutes on days -5 to -3. Patients then receive TriCAR19.20.22 T cells IV over 5-30 minutes on day 0. Patients also undergo echocardiography or MUGA at baseline and blood sample collection and bone marrow biopsy and aspiration throughout the study. Additionally, patients undergo positron emission tomography PET/CT as clinically indicated throughout the study.
  Interventions: Biological: Autologous Anti-CD19/CD20/CD22 CAR T-cells; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Procedure: Echocardiography Test; Drug: Fludarabine; Procedure: Multigated Acquisition Scan; Procedure: Pheresis; Procedure: Positron Emission Tomography
- Cohort B (TriCAR19.20.22 T cells) (Experimental): Patients undergo apheresis between days -30 and -7 or days -9 and -7. Patients receive lymphodepletion chemotherapy with cyclophosphamide IV on day -6, fludarabine IV over 30 minutes on days -5 to -3 and TriCAR19.20.22 T cells IV over 5-30 minutes on days 0 and 7. Patients also undergo echocardiography or MUGA at baseline and blood sample collection and bone marrow biopsy and aspiration throughout the study. Additionally, patients undergo PET/CT as clinically indicated throughout the study.
  Interventions: Biological: Autologous Anti-CD19/CD20/CD22 CAR T-cells; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Procedure: Echocardiography Test; Drug: Fludarabine; Procedure: Multigated Acquisition Scan; Procedure: Pheresis; Procedure: Positron Emission Tomography

INTERVENTIONS:
Biological: Autologous Anti-CD19/CD20/CD22 CAR T-cells — Given IV
  Other Names: Autologous Anti-CD19/CD20/CD22 CAR T Cells; Autologous Anti-CD19/CD20/CD22 CAR-T Cells; Autologous CAR19.20.22 CAR T-cells
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Pheresis — Undergo apheresis
  Other Names: Apheresed; Apheresis; Blood Component Removal; Collection, Apheresis/Leukapheresis; Hemapheresis
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase I trial tests the safety, side effects and best dose of anti-CD19/20/22 chimeric antigen receptor (CAR) T cells (TriCAR19.20.22 T cells) and how well they work in treating patients with non-Hodgkin lymphoma, acute lymphoblastic leukemia (ALL) and chronic lymphocytic leukemia (CLL) that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). CAR T-cell therapy is a type of treatment in which a patient's T cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. T cells are taken from a patient's blood. Then the gene for a special receptor that binds to a certain protein, such as CD19, CD20 and CD22, on the patient's cancer cells is added to the T cells in the laboratory. The special receptor is called a CAR. Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers. Giving TriCAR19.20.22 T cells may be safe, tolerable, and/or effective in treating patients with relapsed or refractory non-Hodgkin lymphoma, ALL and CLL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety of the treatment of relapsed/refractory non-Hodgkin lymphoma, relapsed/refractory chronic lymphocytic leukemia, lymphoid blast crisis from chronic myeloid leukemia and relapsed/refractory acute lymphoblastic leukemia with chimeric antigen receptor T cells targeting CD19/20/22 and to find the recommended phase II dose for this cellular therapy.

SECONDARY OBJECTIVES:

I. To describe the safety profile of the infusion of CAR-T cells targeting CD19/20/22 in relapsed/refractory non-Hodgkin lymphoma, relapsed/refractory chronic lymphocytic leukemia, lymphoid blast crisis from chronic myeloid leukemia and in relapsed/refractory acute lymphoblastic leukemia.

II. To describe the toxicities related to infusion of CAR-T cells targeting CD19/20/22.

III. To describe the overall response rate and complete response rate of relapsed B cell malignancies treated with CAR-T cells targeting CD19/20/22.

IV. To describe the overall and progression free survival of patients with relapsed lymphoma, CLL, and ALL treated with autologous anti-CD19/CD20/CD22 CAR T-cells (TriCAR19.20.22 T cells).

CORRELATIVE OBJECTIVES:

I. To describe the persistence of TriCAR19.20.22 T cells, measured by flow cytometry and quantitative polymerase chain reaction (qPCR).

II. To describe the T cell subpopulations of the TriCAR19.20.22 T cell product before infusion.

III. To describe the changes in TriCAR19.20.22 T cells after infusion and their correlation with disease response and adverse events.

IV. To investigate the correlation between changes in cytokine plasma concentrations and changes in TriCAR19.20.22 T cell subpopulations over time.

V. To investigate proteomic changes in TriCAR19.20.22 T cell subpopulations over time.

VI. To investigate whether antigen escape occurs in patients treated with TriCAR19.20.22.

OUTLINE: This is a dose-escalation study of TriCAR19.20.22 T cells. Patients are assigned to 1 of 2 cohorts.

COHORT A: Patients undergo apheresis between days -30 and -7 or days -9 and -7. Patients receive lymphodepletion chemotherapy with cyclophosphamide intravenously (IV) on day -6, fludarabine IV over 30 minutes on days -5 to -3. Patients then receive TriCAR19.20.22 T cells IV over 5-30 minutes on day 0. Patients also undergo echocardiography or multigated acquisition scan (MUGA) at baseline and blood sample collection and bone marrow biopsy and aspiration throughout the study. Additionally, patients undergo positron emission tomography (PET)/computed tomography (CT) as clinically indicated throughout the study.

COHORT B: Patients undergo apheresis between days -30 and -7 or days -9 and -7. Patients receive lymphodepletion chemotherapy with cyclophosphamide IV on day -6, fludarabine IV over 30 minutes on days -5 to -3 and TriCAR19.20.22 T cells IV over 5-30 minutes on days 0 and 7. Patients also undergo echocardiography or MUGA at baseline and blood sample collection and bone marrow biopsy and aspiration throughout the study. Additionally, patients undergo PET/CT as clinically indicated throughout the study.

After completion of study treatment, patients are followed for up at 7, 14, 21, 30, 60, and 90 days, at 6 and 12 months, then yearly for up to year 15.

ELIGIBILITY:
Inclusion Criteria:

* COHORT A: Subjects must have relapsed or refractory non-Hodgkin lymphoma with lesions ≤ 5 cm, indolent lymphomas, or chronic lymphocytic leukemia without Richter's transformation
* COHORT B: Subjects with lymphoid blast crisis from chronic myeloid leukemia, acute lymphoblastic leukemia, chronic lymphocytic leukemia with Richter's transformation, non-Hodgkin lymphoma with lesions > 5 cm and/or lymphoblastic lymphoma, or non-Hodgkin lymphoma with circulating lymphoma cells
* Subjects must have been treated with at least two lines of therapy; subjects with prior commercial or investigational CAR T therapy targeting CD19, and/or CD20, and/or CD22 are permitted. Disease must have either progressed after the last regimen or presented failure to achieve complete remission with the last regimen
* Note: Cohort assignment at discretion of principal investigator (PI) depending on patient disease/ history
* Subjects with relapsed/refractory CLL after at least 2 prior lines of appropriate therapy and must have previously received an approved Bruton's tyrosine kinase (BTK) inhibitor and venetoclax
* In subjects who had a prior autologous stem cell transplant for refractory high-grade B-cell lymphoma who relapse within 12 months of autologous stem cell transplant are eligible
* Subjects with relapsed/refractory acute B-lymphoblastic leukemia who received at least 2 prior lines of appropriate therapy. Subjects are also eligible if they have failed or are ineligible for allogeneic stem cell transplant
* Subjects with relapsed/refractory lymphoid blast crisis from prior chronic myeloid leukemia (CML) who received at least 2 prior lines of therapy (tyrosine kinase inhibitors, multiagent chemotherapy) or have failed or are ineligible for allogeneic stem cell transplant
* The patient's lymphoid malignancy must be positive for CD19 and/or CD20 and/or CD22, either by immunohistochemistry or flow cytometry analysis on the last biopsy available or peripheral blood for circulating disease
* Subjects with prior commercial or investigational CAR T therapy targeting CD19, and/or CD20, and/or CD22 are permitted if it has been at least 30 days since previous CAR T cell therapy and < 5% of circulating levels of CD3+ cells express the prior CAR by flow cytometry
* Subjects who received antibodies targeting CD19, or CD20, or CD22 are eligible
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Total bilirubin ≤ 1.5 times the institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) ≥ 3 x institutional upper limit of normal
* Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x institutional upper limit of normal
* Creatinine clearance more than or equal to 50 ml/min calculated by the Cockcroft-Gault formula
* Subjects must have adequate pulmonary function as defined as pulse oximetry ≥ 92% on room air
* Subjects must have adequate cardiac function as defined as left ventricular ejection fraction ≥ 40% in the most recent echocardiogram
* Absolute lymphocyte count ≥ 100/uL; if white blood cell (WBC) is low and differential is not performed, CD3 count (helper/suppressor) should be ≥ 100/ul
* Subjects (or legal guardians) must have the ability to understand and the willingness to sign a written informed consent document
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 6 months after the TriCAR19.20.22 T cell infusion

  * A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (< 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus)
  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptive s that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception
* For men: Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

  * With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 6 months after the TriCAR19.20.22 T cell infusion. Men must refrain from donating sperm during this same period
  * With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 6 months after the TriCAR19.20.22 T cell infusion to avoid potential embryonal or fetal exposure. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception

Exclusion Criteria:

* Autologous transplant within 6 weeks of planned CAR-T cell infusion
* Allogeneic stem cell transplant or donor lymphocyte infusion within 2 months of planned CAR-T cell infusion and patients must be off immunosuppressive agents
* Subjects with live vaccines given 28 days prior to lymphodepleting (LD) chemotherapy will be excluded
* Active graft versus host disease
* Active central nervous system or meningeal involvement by lymphoma or leukemia
* Subjects with untreated brain metastases/central nervous system (CNS) disease will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Subjects with a history of CNS or meningeal involvement must be in a documented remission by cerebrospinal fluid (CSF) evaluation and contrast- enhanced magnetic resonance imaging (MRI) imaging for at least 90 days prior to registration
* Active malignancy, other than non-melanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast). Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial (e.g. low Gleason score prostate cancer)
* A minimum of 28 days must have elapsed between prior treatment with investigational agent(s) and the day of lymphocyte collection
* HIV-seropositive patients are allowable, however must be on effective anti-retroviral therapy with undetectable viral load within 6 months of enrollment to be eligible for this trial
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, pulmonary abnormalities or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breastfeeding women are excluded from this study because CAR-T cell therapy may be associated with the potential for teratogenic or abortifacient effects. Women of childbearing potential must have a negative serum pregnancy test. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with CAR-T cells, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study
* Evidence of myelodysplasia or cytogenetic abnormality indicative of myelodysplasia on any bone marrow biopsy prior to initiation of therapy
* Subjects with a positive hepatitis B core antibody or surface antigen are at high risk for hepatitis B virus (HBV) reaction and will require entecavir/tenofivir prophylaxis or serial hepatitis B (Hep) B polymerase chain reaction (PCR) monitoring at the direction of an infectious disease specialist. Duration of prophylaxis to correspond with detection of TriCAR19.20.22 T cells/viral vector copies in serum or continued evidence of B-cell aplasia such as reduced intravenous immunoglobulin (IVIG) levels. No antiviral prophylaxis is indicated with hepatitis C positivity with negative PCR
* Subjects with history of clinically relevant CNS pathology such as epilepsy, seizure disorders, paresis, aphasia, uncontrolled cerebrovascular disease, severe brain injuries, dementia and Parkinson's disease
* History of autoimmune disease (i.e. rheumatoid arthritis, systemic lupus erythematosus) with requirement of immunosuppressive medication within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Up to 30 days after infusion
  Adverse events will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 with the exception of cytokine release syndrome (CRS). CRS will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) Consensus Grading for CRS.
Recommended phase 2 dose | Up to 30 days after infusion

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days after infusion
  Will be described and graded according to NCI CTCAE v 5.0. CRS will be described and graded using ASTCT Consensus Grading for CRS. Will be evaluated with descriptive statistics for the frequencies of AEs of different grades.
Overall response rate | Up to 15 years
  Will be evaluated with proportions used to describe response rates.
Complete response rate | Up to 15 years
  Will be evaluated with proportions used to describe response rates.
Overall survival | Up to 15 years
  Will be calculated using Kaplan-Meier method, comparisons between groups will be done using the log rank test.
Progression-free survival | From entry onto study until lymphoma progression or death from any cause, assessed up to 15 years
  Will be calculated using Kaplan-Meier method, comparisons between groups will be done using the log rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Sumithira Vasu, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu